CLINICAL TRIAL: NCT03245294
Title: Analysis of Factors Contributing to the Pressure Wave Form Changes During Lumbar Epidural Injections
Brief Title: Factors Contributing to the Pressure Wave Form Changes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, Ji Hee Hong, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2017-05-039
Record Dates: First submitted 2017-08-03; First posted 2017-08-10 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Analysis, Event History
Keywords: cervical epidural space; abrupt pressure decrease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumbar ESI with paramedian approach (Active Comparator): Lumbar ESI with paramedian approach
  Interventions: Procedure: lumbar epidural injection
- Lumbar ESI with midline approach (Active Comparator): Lumbar ESI with midline approach
  Interventions: Procedure: lumbar epidural injection

INTERVENTIONS:
Procedure: lumbar epidural injection — the pattern of pressure decrease from ligamentum flavum to epidural space

SUMMARY:
The purpose of this study is to evaluate the decrease pattern of lumbar epidural pressure from ligamentum flavum to epidural space and analyzing factors contributing this pressure change pattern.

DETAILED DESCRIPTION:
Loss of resistance (LOR) is the most commonly used method to confirm the epidural space. The advantage of LOR is its simplicity; only saline or air filled syringe is required. LOR is felt through the sudden decrease of pressure and this pressure gradient is generated when the needle is within the passage of interspinous ligament, ligamentum flavum and epidural space. The presence of ligamentum flavum is crucial for the identification of epidural space by LOR. However, gaps in ligamentum flavum, paravertebral muscle and cyst in interspinous ligament can modify this passage and a false LOR is generated consequentially. The false positive rate of the lumbar and cervical area was reported to be 8.3~17% and 30~68%, respectively. If the false positive rate is high, repeated attempts of epidural steroid injection (ESI) are required, with additional discomfort or pain to the patient.

The high rate of false LOR has prompted the design of adjunctive modalities. Among these, epidural pressure waveform analysis (EPWA) using pressure transducer has been reported. If the epidural needle or catheter is positioned accurately in the epidural space, a pulsatile wave coinciding with arterial pulsations can be seen through the monitor.

Recent study suggested that significant abrupt pressure decrease occurs when cervical epidural injection was done via paramedian approach rather than midline.

ELIGIBILITY:
Inclusion Criteria:

* lumbar herniated nucleus
* lumbar spinal stenosis
* internal disc disruption
* NRS > 5
* ODI > 20

Exclusion Criteria:

* coagulopathy
* allergy to contrast media
* infection at needle insertion site
* absence of lumbar MRI
* Pregnancy
* previous lumbar spine surgery
* neurological symptoms requiring prompt reevalution

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
pattern of epidural pressure decrease | 1 second after the completion of entry from ligamentum flavum to epidural space
  abrupt or gradual decrease of epidural pressure

SECONDARY OUTCOMES:
factors contributing the epidural pressure pattern | 60 minutes after the completion of entry from ligamentum flavum to epidural space
  factors contributing the epidural pressure decrease(abrupt vs. gradual) pattern

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hee Hong, PhD, Principal Investigator — Keimyung University
Locations (1):
- Ji Hee Hong, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No